CLINICAL TRIAL: NCT03499756
Title: A Couple-based Interpersonal Psychotherapy on Postnatal Depression and Family Sense of Coherence: a Randomized Controlled Trial
Brief Title: Couple-based Interpersonal Psychotherapy on Postnatal Depression and Family Sense of Coherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Ngai Fei Wan, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PolyU 156082/17H
Record Dates: First submitted 2018-04-03; First posted 2018-04-17 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Postnatal Depression
Keywords: Postnatal depression, interpersonal psychotherapy
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Couple-based interpersonal psychotherapy (Experimental): The intervention consists of three weekly 2-hour antenatal sessions and two 30-minute telephone follow-up sessions delivered within four weeks postpartum.
  Interventions: Behavioral: Couple-based interpersonal psychotherapy
- Control (No Intervention): The control group will receive the standard prenatal and postnatal care.

INTERVENTIONS:
Behavioral: Couple-based interpersonal psychotherapy — The contents include: (1) an overview of changes associated with the role transition of parenthood and an introduction to the coping skills relating to role transition and parenting; (2) discussing common postpartum and interpersonal difficulties, such as conflicts with partners or extended family, and teaching effective communication skills to resolve interpersonal conflicts and maintain a good interpersonal relationship; and (3) building family strengths and resources by enhancing family sense of coherence, such as reassessing the challenges of the new role, applying problem solving techniques to deal with role transition and interpersonal problems, and developing new social support.
  Arms: Couple-based interpersonal psychotherapy

SUMMARY:
Postnatal depression is a common public health problem which has long-term sequelae on the family and the infant's psychosocial development. Interpersonal psychotherapy has demonstrated its value as one of the most effective interventions for postnatal depression. The aim of this study is to examine the effect of a couple-based interpersonal psychotherapy for first-time Chinese mothers and fathers on depressive symptoms, family sense of coherence, and marital relationships immediately after intervention and at 6 weeks and 6 months postpartum.

DETAILED DESCRIPTION:
Background: Postnatal depression is a common public health problem which has long-term sequelae on the family and the infant's psychosocial development. Interpersonal psychotherapy has demonstrated its value as one of the most effective interventions for postnatal depression. Enhancement of family sense of coherence may be helpful for women who are at risk for postnatal depression. However, few studies in the context of Chinese parenthood have evaluated the effect of interpersonal psychotherapy on postnatal depression and the underlying mechanisms.

Aim: To examine the effect of a couple-based interpersonal psychotherapy for first-time Chinese mothers and fathers on depressive symptoms (primary outcome), family sense of coherence (secondary outcome), and marital relationships (secondary outcome) immediately after intervention and at 6 weeks and 6 months postpartum.

Method: A randomized controlled trial will be used to evaluate the effect of a couple-based interpersonal psychotherapy on depressive symptoms (primary outcome), family sense of coherence (secondary outcome), and marital relationships (secondary outcome) immediately after intervention and at 6 weeks and 6 months postpartum. A convenience sample of 125 couples will be recruited at the antenatal clinics and randomly assigned to either experimental or control group. The experimental group will receive the intervention in addition to the standard perinatal care, while the control group will only receive the standard perinatal care.

Intervention: The intervention consists of three weekly 2-hour antenatal sessions using an interpersonal psychotherapy approach that focused on enhancement of family sense of coherence and two telephone follow-ups within the first four weeks after delivery.

Outcome measures: The primary outcome measure of postnatal depression will be assessed by the Edinburgh Postnatal Depression Scale. Secondary outcome measures of family sense of coherence and the marital relationship, will be assessed by the Family Sense of Coherence Scale and Dyadic Adjustment, respectively, at baseline, immediately post-intervention, 6 weeks and 6 months postpartum.

Data analysis: Linear mixed models will be used to test for significant differences between the groups on outcome variables.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or above;
* married, first-time parents, live together;
* able to speak and read Chinese; and Hong Kong residents.

Exclusion Criteria:

* a present history of psychiatric illness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 455 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale | 6 weeks postpartum
  Edinburgh Postnatal Depression Scale is a 10-item self-report scale assessing the presence of depressive symptoms in the postnatal period. Each item is scored on a 4-point scale with total scores ranging from 0 to 30. Higher score indicates greater depressive symptoms, i.e. worse outcome.

SECONDARY OUTCOMES:
Edinburgh Postnatal Depression Scale | 6 months postpartum
  Edinburgh Postnatal Depression Scale is a 10-item self-report scale assessing the presence of depressive symptoms in the postnatal period. Each item is scored on a 4-point scale with total scores ranging from 0 to 30. Higher score indicates greater depressive symptoms, i.e. worse outcome.
Family Sense of Coherence Scale (Short Form) | 6 weeks postpartum
  Family Sense of Coherence Scale Short Form is a 12-item scale assessing the extent to which the family perceives the environment as meaningful, comprehensible and manageable. Each item is scored on a 7-point scale, with total scores ranging from 7 to 84. Higher scores indicates a stronger perception of family life coherence, i.e. better outcome.
Family Sense of Coherence Scale (Short Form) | 6 months postpartum
  Family Sense of Coherence Scale Short Form is a 12-item scale assessing the extent to which the family perceives the environment as meaningful, comprehensible and manageable. Each item is scored on a 7-point scale, with total scores ranging from 7 to 84. Higher scores indicates a stronger perception of family life coherence, i.e. better outcome.
Dyadic Adjustment Scale | 6 weeks postpartum
  Dyadic Adjustment Scale is a 32-item measure with four sub-scales: consensus (13 items), satisfaction (10 items), cohesion (5 items), and affectional expression (4 items). A total score is calculated by summing all four subscales' score, with a range of 0-151. Higher scores indicates better adjustment to one's relationship, i.e. better outcome.
Dyadic Adjustment Scale | 6 months postpartum
  Dyadic Adjustment Scale is a 32-item measure with four sub-scales: consensus (13 items), satisfaction (10 items), cohesion (5 items), and affectional expression (4 items). A total score is calculated by summing all four subscales' score, with a range of 0-151. Higher scores indicates better adjustment to one's relationship, i.e. better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Elizabeth Hospital, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No